CLINICAL TRIAL: NCT00934960
Title: Distance, Intermediate and Near Visual Outcomes, Range of Vision and Patient Satisfaction After Bilateral Implantation of Different Multifocal IOLs
Brief Title: Multifocals and Accommodating/Bilateral Implantation of Different Multifocal Intraocular Lens (IOLs)
Status: Terminated | Type: Observational
Why Stopped: PI separated employment from the university.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Dr. Helga Sandoval/Principal Investigator, Medical University of South Carolina
Other Study IDs: MRC 09-001
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Cataracts
Keywords: vision; Intraocular lenses
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate vision at different distances (far (13 ft), intermediate (2.0 ft) and near (13 to 15 in)) with and without the patient's glasses (if the patient wears them), range of vision (the difference between the farthest distance and the closest distance that the patient can comfortably read 20/25 of the near card), and patient satisfaction (how satisfied/happy is the patient with their vision) following bilateral implantation of different multifocal IOLs after routine phacoemulsification.

The patients are being asked to participate in this study because you have had cataract surgery and have received one of the IOLs implanted: ReSTOR +4.0 D, ReSTOR +3.0 D, Crystalens, and/or ReZoom. The investigator in charge of this study is Dr. Helga Sandoval. This study is being conducted at Storm Eye Institute at the Medical University of South Carolina and will involve approximately 50 volunteers.

DETAILED DESCRIPTION:
STUDY DESIGN:

This is a prospective, non-randomized, unmasked pilot study.

1. SETTING:

   Storm Eye Institute, Medical University of South Carolina, Charleston, SC
2. SUBJECTS

A total of 50 patients of both sexes and any race or ethnic background who underwent uneventful routine bilateral cataract extraction and multifocal or accommodating intraocular lens implantation will be included. Subjects will be divided in 5 groups of 10 subjects each based on the IOL implanted as follows: ReSTOR +4.0 D, ReSTOR +3.0 D, Crystalens, ReZoom, and Mix-and-match (patients implanted with ReSTOR in one eye and ReZoom in the fellow eye).

Assessment included a thorough medical history and a complete eye examination. The latter will include ETDRS visual acuity at distance (4 mts), intermediate (60 cm) and near (33 or 40 cm accordingly to the lens, under photopic conditions) evaluated uncorrected and best-corrected as well as distance-corrected near and intermediate visual acuity, , and range of vision (uncorrected and distance-corrected); the previous tests will be done per eye and both eyes (visual summation). Slit-lamp exam, eye dominance, stereopsis, pupil size under photopic conditions, corneal topography and a satisfaction questionnaire will be evaluated as well. A defocus curve will be performed as follows: a phoropter and a 100% contrast ETDRS chart positioned 4 meters from the subject under photopic lighting conditions will be used. Manifest refraction will be used to designate the zero (0) baseline. To begin the testing, subjects will be defocused -5.00 D spherical correction from their best distance correction (manifest refraction). The logMAR acuity at this refraction will be recorded. Minus spherical power will be decreased in 0.50 D increments (i.e., -4.50 D, -4.00 D, -3.50 D, etc.) with logMAR acuity recorded at each change in correction until only the best distance correction (manifest refraction) remains. In a further step, subjects will be defocused +2.00 D spherical correction from the best distance correction (manifest refraction) and the logMAR acuity will be recorded. Plus spherical power will be decreased in 0.50 D increments (i.e., +1.50 D, +1.00 D, +0.50 D) with logMAR acuity recorded at each change in correction until only the best distance correction (manifest refraction) remains.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST fulfill the following conditions to qualify for enrollment into the trial

* Subject must have a multifocal or an accommodating IOL implanted bilaterally.
* Age: 40 to 90 years old.
* At least 3 months after cataract extraction and intraocular lens implantation in the second eye.
* Willing and able to comply with scheduled visit and other study procedures.

Exclusion Criteria:

Subjects with ANY of the following conditions on the eligibility exam may NOT be enrolled into the trial.

* Ocular pathology affecting visual acuity: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmus or macrophthalmus, optic nerve atrophy, macular degeneration (with best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Keratometric astigmatism exceeding 2.00 diopters.
* Planned postoperative refraction for mono-vision.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in either eye.
* Other ocular surgery at the time of the cataract extraction.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients of both sexes and any race or ethnic background who underwent uneventful routine bilateral cataract extraction and multifocal or accomodating intraocular lens implantation will be included. Subjects will be divided in 5 groups of 10 subjects each based on the IOL implanted as follows: ReSTOR +4.0 D, ReSTOR +3.0 D, Crystalens, ReZoom, and Mix-and-match (patients implanted with ReSTOR in one eye and ReZoom in the fellow eye).
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate visual outcomes at distance, intermediate and near as well as range of vision and patient satisfaction after bilateral implantation of multifocal or accommodating IOLs post routine cataract extraction at least 3 months after surgery. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Helga P Sandoval, MD, Principal Investigator — Associate Professor
Locations (1):
- Helga Sandoval, MD, Charleston, South Carolina, United States